CLINICAL TRIAL: NCT04344431
Title: Management by Hyperbaric Oxygen Therapy of Patients With Hypoxaemic Pneumonia With SARS-CoV-2 (COVID-19)
Acronym: OHB10cov
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020PPRC03
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Covid-19
Keywords: Sars-CoV2; Pneumonia; Hypoxaemic; Oxygen-dependence; Hyperbaric oxygen; Respiratory decompensation
MeSH Terms: conditions — COVID-19; Pneumonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBO group (Experimental)
  Interventions: Combination Product: Hyperbaric oxygen treatment (HBOT) i.e. inhalation of pressurized oxygen delivered by a hyperbaric chamber (drug/device)
- Non-HBO group (No Intervention)

INTERVENTIONS:
Combination Product: Hyperbaric oxygen treatment (HBOT) i.e. inhalation of pressurized oxygen delivered by a hyperbaric chamber (drug/device) — One session per day of HBOT in addition to the standard treatment with normobaric oxygen
  Arms: HBO group

SUMMARY:
Several patients with hypoxaemic SARS-CoV2 pneumonia were able to benefit from hyperbaric oxygen treatment (HBOT) in China. In a clinical case published in the Chinese journal of hyperbaric medicine, treatment with repeated HBO sessions prevented admission to intensive care unit with mechanical ventilation in a patient aged 69 who presented with signs of respiratory decompensation. HBOT is the most powerful oxygenation modality in the body today. HBOT can dramatically increase the amount of dissolved oxygen in the blood. HBOT not only promotes blood transport but also its tissue delivery. Furthermore, HBOT has specific immunomodulatory properties, both humoral and cellular, making it possible, for example, to reduce the intensity of the inflammatory response and to stimulate antioxidant defenses by repeating sessions. A virucidal capacity of HBOT might also be involved. HBOT is generally regarded as safe with very few adverse events.

Following this feedback, it is proposed in the context of crisis management related to SARS-CoV2 to assess the value of HBO treatment of patients with CoV2 pneumonia. Indeed, it seems essential to propose therapeutic strategies to limit the risk of respiratory decompensation requiring admission to intensive care unit for patients with SARS-CoV2 pneumonia.

DETAILED DESCRIPTION:
The main objective of this study is to assess the effectiveness of HBOT in addition to normal management over the period of normalization of the oxygen requirement (oxygen dependence) in patients with SAR-CoV2 pneumonia not requiring invasive or non-invasive ventilation. It is a prospective, interventional, multicentre, controlled, randomized study. Patients admitted for SARS-CoV2 pneumonia in the Covid sector of the hospital, who have oxygen-dependence criteria will be proposed for inclusion in accordance with the inclusion and non-inclusion criteria. Randomization will be carried out to determine the allocation in two groups: an HBO group which will perform a daily session after checking for the absence of contraindication to HBO and a non-HBO control group with the same clinical criteria, but who will not benefit from HBOT sessions. In both groups, the standard continuous treatment with normobaric oxygen will be maintained.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, Age ≥ 18 years
* Patient with oxygen dependence criterion: need to maintain an oxygen flow rate less than or equal to 6 liters / min to obtain: saturation by pulse oximetry (SpO2) greater than or equal to 92% or arterial gas with value PaO2 greater than 60mmHg.
* Diagnostic confirmation of SARS-CoV-2 pneumonia

Exclusion Criteria:

* Minor subject (age <18 years)
* Person unable to give consent
* Refusal to participate
* Pregnancy
* Participating in another research
* Signs of respiratory decompensation requiring mechanical ventilation
* Diagnosis of pneumonia with SARS-CoV-2 not confirmed
* Oxygen dependence criterion exceeded i.e. need to maintain an oxygen flow rate greater than or equal to 6 liters / min to obtain: saturation by pulse oximetry (SpO2) greater than or equal to 92% or arterial gas with value of PaO2 greater than 60mmHg.
* Inability to maintain the prolonged sitting position (at least 2 hours)
* Subject with contraindications to HBOT

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-14 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Time to normalize the oxygen requirement (oxygeno-dependence) | 1 month
  Time to normalize the oxygen requirement (oxygeno-dependence), i.e. allowing a pulse oximetry value in ambient air greater than or equal to 92% and / or arterial blood gas with a PaO2 value greater than 60mmHg in ambient air.

SECONDARY OUTCOMES:
Days of hospitalization between the HBO group and the control group. | 1 month
  Number of days with oxygen need, taking into account the predictors of bad outcome
Oxygen flow values to obtain a saturation by pulse oximetry greater than or equal to 92% values between the HBO group and the control group. | 1 month
  Oxygen flow values to obtain a saturation by pulse oximetry greater than or equal to 92% between the OHB group and the control group.
Days on invasive mechanical ventilation | 1 month
  Days on invasive mechanical ventilation
Mortality | 1 month
  Mortality

OTHER OUTCOMES:
Number of patients requiring a permanent O2 flow rate greater than 6 liters / min with high-speed nasal mask or oxygen therapy or with invasive or non-invasive ventilation | 1 month
  Number of patients requiring a permanent O2 flow rate greater than 6 liters / min with high-speed nasal mask or oxygen therapy or with invasive or non-invasive ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Eric BLATTEAU, MD, PhD, Principal Investigator — Sainte-Anne military hospital
Locations (3):
- France (3):
  - Hôpital d'Instruction des Armées Laveran, Marseille
  - Centre Hospitalier Intercommunal de Toulon - La Seyne-sur-Mer, Toulon
  - Hôpital d'Instruction des Armées Sainte-Anne, Toulon

IPD SHARING:
Plan to Share IPD: No